CLINICAL TRIAL: NCT07402746
Title: Sensorimotor Training to Enhance Performance - the STEP AHEAD Program
Acronym: STEP AHEAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sport Injury Prevention Research Centre (Other)
Responsible Party: Principal Investigator, KSchneider, Associate Professor, Clinician Scientist (Physiotherapist), Sport Injury Prevention Research Centre
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: STEP AHEAD
Record Dates: First submitted 2024-07-24; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Ice Hockey Players
Keywords: training; Sensorimotor; Neuromuscular; Prevention

STUDY DESIGN:
Intervention Model Description: Initial control intervention for four weeks of typical off season training followed by a second step where the sensorimotor and neuromuscular training is introduced.
Masking Description: Due to the nature of the trial it is not possible to mask the participants or the outcome assessors. However, the outcome assessors and participants will be blinded to the previous scores on the outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sensorimotor and neuromuscular training (Experimental): Sensorimotor and neuromuscular training added in addition to typical off season ice hockey training as outlined in the typical training arm.
  Interventions: Other: sensorimotor and neuromuscular training; Other: Typical off season ice hockey training
- Typical off season training (Active Comparator): Typical of season training includes strength and conditioning, ice hockey on ice drills as per the Crash Conditioning typical training.
  Interventions: Other: Typical off season ice hockey training

INTERVENTIONS:
Other: sensorimotor and neuromuscular training — Sensorimotor and neuromuscular training exercises aimed at training the cervical spine neuromuscular control, vestibular system and oculomotor system in addition to ice hockey specific training the incorporates higher level integrated functional activities of these integrated systems. This will be performed at the same frequency as their typical training - four days per week in the gym, one day of yoga or recovery as well as on ice sessions.
  Arms: Sensorimotor and neuromuscular training
Other: Typical off season ice hockey training — Typical training for ice hockey players off season

SUMMARY:
The goal of this study is to evaluate the effects of SM/NM training in ice hockey players. The specific questions include: 1) typical performance on sensorimotor and neuromuscular (SM/NM) tests 2) evaluate SM/NM training on ice hockey skills performance and SM/NM tests, 3) evaluate SM/NM control to prevent concussions and injuries

Participants will:

Consent and complete a series of SM/NM tests. Participate in their typical training for 4 weeks. Repeat the SM/NM tests. Participate in SM/NM training for 4 weeks as part of their off season training program.

Repeat the SM/NM tests and on ice skills testing. Record any injuries and concussions that they sustain over the next season. Repeat the SM/NM tests and on ice skills tests at the start of the 2025 off season training (estimated May - July of 2025).

DETAILED DESCRIPTION:
Rationale:

While sensorimotor function is recognized as an important aspect of growth and development, little is known about specific changes in sensorimotor control with sport specific training. Similarly, the relationship between sensorimotor control and sport-specific performance is not yet well understood. Specific rehabilitation exercises have been shown to improve sensorimotor control, many of which are context specific and may also prevent injury and/or concussion. The effect of age on these outcomes and the relationship between training sensorimotor control and age is also not well understood. Thus, evaluation of sensorimotor control outcomes across ages, the effects of sensorimotor training on sensorimotor control and performance is needed and may inform changes to recommendations for sport-specific training.

Ultimately, understanding the effect of training specific sensorimotor systems (which is not a part of typical sport training environments) will inform multiple areas of sport including: 1) Sport-specific performance 2) typical development of SM/NM function, 3) the effect of SM/NM training on SM/NM measures and ice hockey specific physical performance and 4) injury and concussion prevention strategies.

Therefore, the objectives of this study are to:

1. Describe age and sex specific typical scores on sensorimotor and neuromuscular (proprioception, movement related, balance, vision, divided attention) and ice hockey specific physical performance measures over one off season of training.
2. Evaluate the effects of a sensorimotor training program on ice hockey skills performance.
3. Evaluate sensorimotor control as a means to improve safety in sport:

   1. Evaluate the effect of SM/NM training on concussion and injury risk.
   2. Evaluate the effect of previous concussion and injury on sensorimotor function.
4. Evaluate the effect of SM/NM training on performance of 1) system specific outcomes and 2) sport specific measures in ice hockey players.

ELIGIBILITY:
Inclusion Criteria:Ice hockey players in Calgary and area who are training with Crash Conditioning for the 2024-2026 off season -

Exclusion Criteria:

N/A

-

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-05-18 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Craniocervical flexion | 0 weeks, 4 weeks, 8 weeks each year, up to 2 years
  mmHg, the ability of the participant to perform a craniovertebral flexion task in a controlled way and maintain the position for a minimum of 3 seconds.
Dynamic Visual Acuity | 0 weeks, 4 weeks, 8 weeks each year, up to 2 years
  logMAR, Represents the ability of the patient to see clearly with head motion as per Schneider et al 2019=8
Vestibular Ocular Motor Screen (VOMS) | 0 weeks, 4 weeks, 8 weeks each year, up to 2 years
  Symptom provocation on tests of vestibulo ocular and oculomotor function, rated on a scale of 0-10 where 0=no symptoms and 10= the worse imaginable, Mucha et al 2014
Advanced Functional Gait Assessment | 0 weeks, 4 weeks, 8 weeks each year, up to 2 years
  /48, 16 tests of dynamic balance each rated on a scale of 0-3 with 0 repress unable to complete the task and 3 is able to perfectly complete the task.
Transition Agility Skate | 0 weeks, 4 weeks, 8 weeks each year, up to 2 years
  Seconds, Outcome of the transition agility skate on the Hockey Canada skills test

SECONDARY OUTCOMES:
Cervical spine range of motion | 0 weeks, 4 weeks, 8 weeks each year, up to 2 years
  1=full range of motion, 0=limited range of motion
Anterolateral flexion strength | 0 weeks, 4 weeks, 8 weeks each year, up to 2 years
  kilograms (kg), average of three trials in a rotated position to either the right or left and defined according to the position of the head
cervical flexor endurance test | 0 weeks, 4 weeks, 8 weeks each year, up to 2 years
  Seconds, the length of time the participant can lift the head in craniovertebral flexion
cervical flexion rotation test | 0 weeks, 4 weeks, 8 weeks each year, up to 2 years
  1=positive, 0=negative, a measure of upper cervical spine dysfunction with a positive test suggesting cervicogenic headache, limited range of motion in full flexion by >20 degrees, measured to the right and left
head perturbation test | 0 weeks, 4 weeks, 8 weeks each year, up to 2 years
  0-8/8; ability of the individual to maintain their head in a neutral position when an external force of 5lbs is applied
Head thrust test | 0 weeks, 4 weeks, 8 weeks each year, up to 2 years
  Positive = 1, Negative =0, Ability of the eyes to maintain a fixed position on a target with rapid head motion
Numeric Pain Rating Scale (NPRS) Headache | 0 weeks, 4 weeks, 8 weeks each year, up to 2 years
  Headache 0-10 where 0=no symptoms and 10=worst symptom imaginable
Numeric Dizziness Rating Scale (NDRS) Dizziness | 0 weeks, 4 weeks, 8 weeks each year, up to 2 years
  dizziness 0-10 where 0=no symptoms and 10=worst symptom imaginable
Numeric Pain Rating Scale (NPRS) Neck pain | 0 weeks, 4 weeks, 8 weeks each year, up to 2 years
  neck pain 0-10 where 0=no symptoms and 10=worst symptom imaginable
Concussion | yearly, up to 2 years
  Defined as per the Amsterdam International Consensus on Concussion in Sport

CONTACTS AND LOCATIONS:
Locations (1):
- Concussion Rehabilitation Laboratory, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No